CLINICAL TRIAL: NCT01422785
Title: A Pilot Study to Evaluate the Efficacy of Fixed Dose Combination Clindamycin Phosphate 1.2%/Tretinoin 0.025% Gel Alone Versus Fixed Dose Combination Clindamycin Phosphate 1.2%/Tretinoin 0.025% Gel Plus Benzoyl Peroxide 6% Foaming Cloths in the Treatment of Facial Acne Vulgaris
Brief Title: A Study Comparing Combination Clindamycin Phosphate/Tretinoin Gel Alone Versus With Benzoyl Peroxide Foaming Cloths for Facial Acne
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeichner, Joshua, M.D. (Individual)
Responsible Party: Principal Investigator, Joshua Zeichner, Zeichner, Joshua, M.D., Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 10-1602
Record Dates: First submitted 2011-08-12; First posted 2011-08-24 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate; Tretinoin; Gels; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clindamycin phosphate 1.2%/tretinoin 0.025% gel alone (Active Comparator)
  Interventions: Drug: clindamycin phosphate 1.2%/tretinoin 0.025% gel alone
- clindamycin / tretinoin gel plus benzoyl peroxide (Active Comparator)
  Interventions: Drug: clindamycin phosphate 1.2%/tretinoin 0.025% gel plus benzoyl peroxide 6% foaming cloths

INTERVENTIONS:
Drug: clindamycin phosphate 1.2%/tretinoin 0.025% gel alone — Once daily application of the clindamycin phosphate 1.2%/tretinoin 0.025% gel in the evening
  Arms: clindamycin phosphate 1.2%/tretinoin 0.025% gel alone
Drug: clindamycin phosphate 1.2%/tretinoin 0.025% gel plus benzoyl peroxide 6% foaming cloths — wash face with the benzoyl peroxide foaming cloth then rinse. then apply clindamycin phosphate 1.2%/tretinoin 0.025% gel. both done in the evening.
  Arms: clindamycin / tretinoin gel plus benzoyl peroxide

SUMMARY:
There are many different factors that cause acne. So combination treatment using different medications that can address these different factors is commonly used to treat acne. Fixed-dose combination clindamycin phosphate 1.2% and tretinoin 0.025% gel and benzoyl peroxide 6% foaming cloths are both used to treat acne. This study will evaluate the use of the medications when used together.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 12 years old.
* Subjects must be in good general health as confirmed by medical history and physical examination.
* Females of child-bearing potential must have a negative urine pregnancy test at the baseline visit and agree to use adequate birth control during the study (barrier, oral, injection, intrauterine or abstinence).
* Clear diagnosis of facial acne vulgaris for at least 3 months.
* Subject must have a static Physician's Global Assessment (PGA) of at least 2 (mild severity), but no more than 4.
* Disease must be stable or slowly worsening for more than one week prior to entering the study.
* Subjects or their guardians must be able to read, sign, and date the informed consent, and abide by study restrictions for its duration.

Exclusion Criteria:

* Females who are pregnant, attempting to conceive, or breastfeeding.
* Subjects with known hypersensitivity to study drug.
* Subjects with very severe acne (PGA score of 5)
* Subjects with overt signs of skin atrophy, telangiectasias or other skin findings that would affect efficacy evaluation.
* Subjects with a current active skin malignancy or infection.
* Subjects requiring the use of medications known to alter the course of acne vulgaris during the study treatment.
* Subjects who have received systemic antibiotics within 2 weeks.
* Subjects using systemic corticosteroids or immunosuppressants within 28 days of entering the study.
* Subjects who have received any topical therapies for acne vulgaris within 2 weeks of entering the study.
* Subjects taking birth control pills for less than 3 months or solely for the prevention of acne.
* Subjects who are currently participating in or, within the previous 28 days, have participated in another study for the treatment of acne vulgaris.
* Subjects with clinical conditions that may post a health risk to the subject by being involved in the study or detrimentally affect regular follow-up of the subject.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change in PGA scores of patients using combination clindamycin phosphate 1.2%/tretinoin 0.025% gel with or without benzoyl peroxide 6% foaming cloths for facial acne | Weeks 2, 4, 8, 12
  The primary efficacy endpoint will be "Treatment Success", a static endpoint defined as a score of 0 (clear) to 1 (almost clear) at Week 12 (final study visit) by PGA scoring system.

SECONDARY OUTCOMES:
Change in Postinflammatory hyperpigmentation score at each study visit and from baseline to final visit. | Weeks 2, 4, 8, 12
  Change in PIH score from baseline will be assessed. (based on a 6 point scale)
Total number of adverse events. | Weeks 2, 4, 8, 12
  Safety/drug-tolerance evaluated at each visit (total number of adverse events)
Change in Subject Self Assessment Scoring Scale | Weeks 2, 4, 8, 12
  Patient rates current severity of their acne.
Change in Acne-Specific Quality of Life Questionnaire (Acne-QoL) | Weeks 2, 4, 8, 12
  Acne-QoL as completed by patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Mt Sinai Hospital - Dept of Dermatology, New York, New York, United States